CLINICAL TRIAL: NCT05046769
Title: COVID-19: A Scope Research on Epidemiology and Clinical Course
Acronym: COVID-Scope
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Saude Publica da Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other); IPATIMUP - Instituto De Patologia E Imunologia Molecular Da Universidade Do Porto (Other)
Responsible Party: Principal Investigator, Margarida Fernandes Tavares, Senior researcher, Instituto de Saude Publica da Universidade do Porto
Other Study IDs: 102-20
Record Dates: First submitted 2021-09-05; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Covid19; SARS CoV 2 Infection; Sequelae of; Infection
Keywords: Covid19; Cohort Studies; Long COVID; Secondary Attack Rate; Serology; Epidemiology
MeSH Terms: conditions — COVID-19; Infections; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe Acute Respiratory Syndrome (SARS) Coronavirus (CoV) 2 infection and the associated coronavirus disease 2019 (COVID-19) are the most recent international health threat challenging our ability to protect populations, to avoid severe outcomes and to understand both the population dynamics of this new condition and the breath of individual responses. Gathering information on the clinical course of the disease and the risk of transmission is essential to design effective therapeutic solutions and preventive measures. The aim of the study proposed, to be carried out at University Hospital Center of "São João" (CHUSJ), is to recruit and follow-up a cohort of patients diagnosed with SARS-CoV-2 infection, to evaluate the clinical course of SARS-CoV-2 infection and COVID-19 cases, to identify prognostic factors and to measure the risk of reinfection. Additionally, researchers intend to characterize the patients and household contacts to describe the dynamics of infection, to calculate household infection attack rate, and to perform the genetic sequencing of SARS-CoV-2 to understand determinants of disease course (namely long-term effects) and risk of household transmission. A sample of participants, identified during the process of evaluation of symptomatic individuals, at the same institution, and negative for SARS-CoV-2 will be selected as negative controls.

Participants will be consecutively recruited and the study is expected to enroll patients as long as the pandemic remains. Information will be gathered based on clinical individual charts, hospital data-bases (example: for administrative data) and individual computer assisted interviews to be performed at pre-defined intervals (3, 12 and 24 months) or according to clinical needs.

The project was approved by the local Ethical Committee and the Data Protection relevant authorities.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with SARS-2-CoV-2 infection treated at CHUSJ and cohabitants able to give informed consent;
* individuals who underwent the test for diagnosis of infection by SARS-CoV-2 at CHUSJ with negative result able to give informed consent.

Exclusion Criteria:

* Inability to obtain informed consent;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with SARS-CoV-2 infection diagnosed at Centro Hospitalar Universitário São João, a level III hospital center, from March 1, 2020. A sample of individuals who underwent the test for diagnosis of infection by SARS-CoV-2 with negative result.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical, biological, psychosocial characteristics | 24 months
  Describe the clinical, biological and psychosocial characteristics SARS-CoV-2 infected inpatients or outpatients identified in our hospital center

SECONDARY OUTCOMES:
Household contacts infection attack rate | 3 months
  Characterize the dynamics of infection
Genome sequence of SARS-CoV-2 | 24 months
  Identify variants of SARS-CoV-2
Reinfection rate | 24 months
  Number and characteristics of reinfections
Prognostic factors of course of disease | 24 months
  Identify clinical, biological and social associated with course of disease

CONTACTS AND LOCATIONS:
Overall Officials: Margarida Tavares, MD, MPH, Principal Investigator — Centro Hospitalar Universitário São João & ISPUP
Locations (1):
- Centro Hospitalar De São João, Porto, Portugal